CLINICAL TRIAL: NCT03426696
Title: Psychological Status and Related Factors of Thyroid Related Eye Disease
Status: Completed | Type: Observational
Sponsor: Huijing Ye (Other)
Responsible Party: Sponsor-Investigator, Huijing Ye, Principal Investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 201701
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Thyroid Related Eye Disease
Keywords: psychological status; Related Factors; Thyroid Related Eye Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid Related Eye Disease: Survey about the psychological condition would done with the patients of Thyroid Related Eye Disease
  Interventions: Behavioral: psychological condition

INTERVENTIONS:
Behavioral: psychological condition — Graves ́ ophthalmopathy quality of life questionnaire, Symptom checklist 90(SLC-90), Hamilton anxiety scale(HAMA), Somatic self-rating scale(SSS), MATRICS Consensus Cognitive Battery (MCCB), Hamilton depression scale(HAMD)

SUMMARY:
The purpose of this study is to evaluate the psychological status of Thyroid Related Eye Disease.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the psychological status of patients of Thyroid Related Eye Disease over 16 years old, and to analyze the related factors of them.

ELIGIBILITY:
Inclusion Criteria:

* over 16 years old
* diagnosed as Thyroid Related Eye Disease

Exclusion Criteria:

* any uncontrolled clinical problems

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients in Sun Yat-sen University that diagnosed as Thyroid Related Eye Disease
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire of patients of Thyroid Related Eye Disease | immediately
  Graves ́ ophthalmopathy quality of life questionnaire (GO-QoL) , The GO-QoL contains 8 questions on visual functioning and 8 questions on appearance; answers on each subscale are transformed to scores ranging from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Symptom checklist 90(SLC-90) | immediately
  It consists of 90 items yielding nine scores along primary symptom dimensions and three scores among global distress indices. The primary symptom dimensions that are assessed are somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and a category of "additional items" which helps clinicians assess other aspect of the clients symptoms. Positive standard includes: total score 160 points or more, or positive items > 43 points, or any item > 2 points.
Hamilton anxiety scale(HAMA) | immediately
  This scale includes 14 items. All projects rated as: asymptomatic, light, medium, heavy, or very heavy. If the total score more than 29 points, there could be severe anxiety; more than 21 points, affirmation have obvious anxiety; more than 14 points, there must be some anxious; more than 7 points might be anxious; if less than 6 points, patients without anxiety symptoms.
Somatic self-rating scale(SSS) | immediately
  Somatic self-rating scale can let the doctor fully understand patients' mood and somatization symptoms. If the selected items scores more than 30 points, the patient may need to clinic treatment.
Hamilton depression scale(HAMD) | immediately
  It is the most common depression clinical application scale. Lower score presents lighter condition, and if the illness is heavier, the higher is the score. There is no depression symptoms for score less than eight points.
Young manic rating scale(YMRS) | immediately
  The Young Mania Rating Scale (YMRS) is a diagnostic questionnaire commonly used to evaluate manic symptoms in patients with bipolar 1 disorder and to assess treatment efficacy in clinical trials. This rating scale comprises eleven items (elevated mood, increased motor activity - energy, sexual interest, sleep, irritability, speech - rate and amount, language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight). The total YMRS score is calculated as the summation of each of the eleven individual item scores.Lower score presents lighter condition, and if the illness is heavier, the higher is the score.There is no manic symptoms for score less than five points.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Ye, Master, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided